CLINICAL TRIAL: NCT06930066
Title: Normal Liver and Spleen Stiffness Values Using Shear Wave Elastography in Children
Brief Title: Normal Pediatric Liver and Spleen SWE
Acronym: SWE
Status: Recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Akif AĞIR, Pediatric Gastroenterologist, Selcuk University
Other Study IDs: 2024/522
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Liver Stiffness; Spleen Stiffness; Shear Wave Elastography in Healthy Children; Normal Organ Elasticity; Pediatric Elastography
Keywords: Shear Wave Elastography; Liver Stiffness; Spleen Stiffness; Pediatric Elastography; Normal Reference Values; Organ Stiffness Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Children: This group includes healthy pediatric participants with no known liver or spleen disease. Each participant will undergo non-invasive shear wave elastography (SWE) to assess liver and spleen stiffness for the purpose of establishing normal reference values.

SUMMARY:
This observational study aims to determine normal liver and spleen stiffness values in healthy children using shear wave elastography (SWE). The study will include participants from the pediatric age group without known liver or spleen disease. SWE measurements will be performed non-invasively to establish reference values. The results may contribute to improving diagnostic accuracy in pediatric elastography applications.

DETAILED DESCRIPTION:
Shear wave elastography (SWE) is a non-invasive imaging method used to assess tissue stiffness. While reference values for SWE have been established in adults, data regarding normal liver and spleen stiffness in children are limited. This single-center, cross-sectional observational study aims to establish normative SWE values for the liver and spleen in the pediatric age group. Children with no known liver or spleen pathology will undergo standardized SWE measurement under controlled conditions. Age-specific and sex-specific reference ranges will be analyzed, which may contribute to enhancing the clinical utility of SWE in pediatric practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 0-18 years
* No known liver or spleen pathology
* Written informed consent obtained from parents or guardians

Exclusion Criteria:

* Known liver disease (e.g., hepatitis, cirrhosis)
* Known spleen disease (e.g., splenomegaly)
* Any history of liver or spleen disease
* Age outside the 0-18 years range

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will consist of healthy children aged 0-18 years, with no known liver or spleen pathology. These participants will be selected from pediatric clinics, specifically those who are seeking routine healthy child check-ups and have no underlying diseases. Non-invasive shear wave elastography (SWE) will be used to assess normal liver and spleen stiffness values. Participants will be selected based on inclusion criteria of being free from any liver or spleen disease, and exclusion criteria will ensure that children with known hepatic or splenic conditions are not included. Parental or guardian consent will be obtained for each participant.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Normal liver and spleen stiffness values | Day 1
  This study aims to establish reference values for liver and spleen stiffness in healthy children using shear wave elastography (SWE).

CONTACTS AND LOCATIONS:
Locations (1):
- Selçuk University Faculty of Medicine, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided